CLINICAL TRIAL: NCT00515502
Title: A Randomised, Double Blind, Placebo-controlled, Double Dummy, 4-way Cross-over, Dose Ascending Study to Assess the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Inhaled Doses of GSK573719 (250, 500 and 1000 μg) and Tiotropium Bromide (18 μg) Via DPI in COPD Patients.
Brief Title: Safety Study Using GSK573719 And Tiotropium In Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AC4108123
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: chronic obstructive pulmonary disease,; GSK573719,; muscarinic receptor antagonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, placebo (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: umeclidinium bromide (UMEC) 250 micrograms (µg), UMEC 500 µg, Tiotropium 18 µg and placebo. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719; Drug: Tiotropium
- Seq 2: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg, placebo (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg and placebo. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719
- Seq 3: UMEC 250 µg, placebo, UMEC 500 µg, UMEC 1000 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: UMEC 250 µg, placebo, UMEC 500 µg and UMEC 1000 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719
- Seq 4: UMEC 250 µg, UMEC 500 µg, placebo, UMEC 1000 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: UMEC 250 µg, UMEC 500 µg, placebo and UMEC 1000 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719
- Seq 5: Placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: Placebo, UMEC 250 µg, UMEC 500 µg and UMEC 1000 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719
- Seq 6: UMEC 250 µg, placebo, Tiotropium 18 µg, UMEC 500 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: UMEC 250 µg, placebo, Tiotropium 18 µg and UMEC 500 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719; Drug: Tiotropium
- Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: Placebo, Tiotropium 18 µg, UMEC 250 µg and UMEC 500 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719; Drug: Tiotropium
- Seq 8: Tiotropium 18 µg, placebo, UMEC 250 µg, UMEC 500 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: Tiotropium 18 µg, placebo, UMEC 250 µg and UMEC 500 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719; Drug: Tiotropium
- Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, placebo (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg and placebo. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719; Drug: Tiotropium
- Seq 10: Tiotropium 18 µg, UMEC 250 µg, placebo, UMEC 500 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: Tiotropium 18 µg, UMEC 250 µg, placebo and UMEC 500 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719; Drug: Tiotropium
- Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: Placebo, UMEC 250 µg, Tiotropium 18 µg and UMEC 500 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719; Drug: Tiotropium
- Seq 12: UMEC 250 µg, placebo, UMEC 500 µg, Tiotropium 18 µg (Active Comparator): Participants received single doses of 4 treatments, over 4 treatment periods, in the following sequence: UMEC 250 µg, placebo, UMEC 500 µg and Tiotropium 18 µg. Treatment periods were seperated by a washout period of at least 14 days.
  Interventions: Drug: GSK573719; Drug: Tiotropium

INTERVENTIONS:
Drug: GSK573719 — 250 micrograms (μg) per blister, administered via dry powder inhaler, dose-ascending study doses began at 250 ug, then 500 ug, and 1000 μg
Drug: Tiotropium — strips of five capsules, each containing 18 μg administered via dry powder inhaler
  Arms: Seq 10: Tiotropium 18 µg, UMEC 250 µg, placebo, UMEC 500 µg; Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg; Seq 12: UMEC 250 µg, placebo, UMEC 500 µg, Tiotropium 18 µg; Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, placebo; Seq 6: UMEC 250 µg, placebo, Tiotropium 18 µg, UMEC 500 µg; Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg; Seq 8: Tiotropium 18 µg, placebo, UMEC 250 µg, UMEC 500 µg; Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, placebo

SUMMARY:
GSK573719 is a high-affinity specific muscarinic receptor (mAChR) antagonist which is being developed for once daily treatment of chronic obstructive pulmonary disease (COPD). The long duration of action of GSK573719 when administered via inhalation in animal models supports the potential for use as a once-daily bronchodilator for COPD.

DETAILED DESCRIPTION:
A randomised, double blind, placebo-controlled, double dummy, 4-way cross-over, dose ascending study to assess the safety, tolerability, pharmacodynamics and pharmacokinetics of single inhaled doses of GSK573719 (3 escalating mcg doses will be used) and tiotropium bromide (18µg) via DPI in COPD patients

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male or female subjects aged 40-75 years inclusive. The need to recruit only Caucasian subjects is related to the need to rigorously exclude 2D6 poor metabolisers based on genotype.
* Female subjects must be of non-childbearing potential.
* An established clinical history of COPD (ATS/ERS definition).
* 'Chronic obstructive pulmonary disease (COPD) is a preventable and treatable disease characterised by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.'
* Subject is a smoker or an ex-smoker with a smoking history of at least 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or equivalent).
* Subject has FEV1/FVC < 0.7 post-bronchodilator (salbutamol) dose.
* Subject has 40 ≥ FEV1 ≤ 80% of predicted normal for height, age and gender after inhalation of salbutamol dose.
* Response to ipratropium bromide.
* Subject is able and has given written informed consent to take part in the study.
* Subject is available to complete all study measurements and procedures.
* Subject's BMI is 18.0 - 32.0 kg/m2.
* Subjects have a 24hr Holter recording that is within normal limits and does not demonstrate any clinically important abnormality that, in the opinion of the investigator, would make the subject unsuitable for participation in the study

Exclusion Criteria:

* Subjects who have a past or present disease of any organ system, which as judged by the Investigator, may affect the outcome of this study.
* The subject has a positive pre-study drug screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cannabis, Cocaine and Opiates. The detection of drugs with a legitimate medical use would not be an exclusion to study participation.
* The subject has a positive pre-study alcohol screen. The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study.
* A suspected history of alcohol abuse within the six months previous to the screening visit.
* The subject has tested positive for hepatitis C antibody, hepatitis B surface antigen or HIV (if determined by local SOP's).
* Subject has received an investigational drug within 30 days of screening.
* The subject is currently taking medication which is known to be a CYP 2D6 inhibitor/substrate.
* The subject has donated a unit (400ml) of blood within 60 days of screening, or, intends to donate during the study.
* The subject has a known allergy or hypersensitivity to ipratropium bromide, tiotropium bromide, atropine and any of its derivatives or lactose/milk protein.
* Subject is unable to use the DISKUS™/HandiHaler devices correctly.
* Subject has prostatic hypertrophy, bladder outlet obstruction, or narrow angle glaucoma.
* Subjects with a 2D6 poor metaboliser genotype (Caucasian).
* The subject has claustrophobia that may be aggravated by entering the plethysmography cabinet (American Association of Respiratory Care 2001 guidelines for body plethysmography)
* Received antibiotic therapy for either a lower respiratory tract infection or for COPD exacerbation within the 4 weeks prior to Screening.

Respiratory criteria

* Subject has a diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, allergic rhinitis, or asthma.
* Subject has poorly controlled COPD, defined as either: acute worsening of COPD that is managed by the subject at home by treatment with corticosteroids in the 6 weeks prior to screening visit Or more than two exacerbations in the previous 6 months prior to screening that required a course of oral corticosteroids or antibiotics, or, for which the subject was hospitalised.
* Subject has participated in a Pulmonary Rehabilitation Program within 4 weeks prior to screening visit or will enter a program during the study.
* Subject has had a respiratory tract infection in the 4 weeks prior to the screening visit.

Cardiovascular criteria

* Current congestive heart failure (greater than NYHA I), myocardial infarction (within 3-years of the screening date) or ischaemic heart disease requiring regular therapy (such as β blockers, long-acting nitrates, calcium antagonists or nicorandil). Aspirin, Clopidogrel and statins are allowed.
* A history of clinically significant arrhythmia or clinically important 24hr Holter findings that, in the opinion of the investigator, would cause a safety concern for entry into the study.
* A mean QTc(B) value at screening >450msec, the QTc(B) of all 3 screening ECGs are not within 10% of the mean, or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T wave)
* Mobitz type II or third degree heart block.
* Risk factors for torsades de pointes (heart failure NYHA II-IV, chronic hypokalaemia, familial long QT syndrome).
* Elevated resting blood pressure or a mean blood pressure equal to or higher than 150/95 mmHg at screening. A history of hypertension is acceptable provided control has been achieved for > 3 months prior to screening with diuretic only.
* A mean heart rate outside the range 50-100 bpm at screening (from vital signs measurement).

Concurrent medication criteria

* Subject requires treatment with inhaled cromolyn sodium or nedocromil, oral β2-agonists, nebulised β2-agonists, nebulised anticholinergics or leukotriene modifiers.
* Subject is unable to abstain from xanthines (other than caffeine) 13-15 days prior to the first dose of study medication until completion of the study (last study-related procedure at the follow-up visit).
* Subject is unable to abstain from short-acting inhaled bronchodilators from 6hrs prior to screening until after completion of screening, or, from 6hrs prior to the administration of study medication until after completion of any given treatment period (i.e. the last assessment in a dosing period).
* Subject is unable to abstain from long-acting inhaled bronchodilators from 72hrs prior to the screening until after completion of all treatment periods (i.e. the last assessment in the final dosing period).
* Subject has changed dose of inhaled corticosteroids within the last 4 weeks, or, will be unable to maintain a constant dose of inhaled corticosteroids during the study.
* Subject is receiving treatment with long term or short-term oxygen therapy or requires nocturnal positive pressure ventilation (CPAP or NIPPV).
* Subject is receiving treatment with beta-blockers, except eye drops, Diltiazem or Verapamil.
* Subject is receiving co-medication with drugs which are commonly recognised to prolong the QTc interval (e.g. quinolones, amiodarone, disopyramide, quinidine, sotalol, chlorpromazine, haloperidol, ketoconazole, terfenadine, cisapride and terodiline).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06-21 (Actual); Primary Completion 2007-11-06 (Actual); Study Completion 2007-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (3):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Tal-Singer R, Cahn A, Mehta R, Preece A, Crater G, Kelleher D, Pouliquen IJ. Initial assessment of single and repeat doses of inhaled umeclidinium in patients with chronic obstructive pulmonary disease: two randomised studies. Eur J Pharmacol. 2013 Feb 15;701(1-3):40-8. doi: 10.1016/j.ejphar.2012.12.019. Epub 2012 Dec 28. PMID 23276660
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: AC4108123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AC4108123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC4108123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC4108123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AC4108123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC4108123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC4108123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive a sequence of 4 of 5 possible treatments over 4 treatment periods each separated by a washout period of at least 14 days. Participants were randomized to receive treatments in 12 possible sequences.
Period: Treatment Period 1
Arm/Group | Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, Placebo | Seq 2: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg, Placebo | Seq 3: UMEC 250 µg, Placebo, UMEC 500 µg, UMEC 1000 µg | Seq 4: UMEC 250 µg, UMEC 500 µg, Placebo, UMEC 1000 µg | Seq 5: Placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg | Seq 6: UMEC 250 µg, Placebo, Tiotropium 18 µg, UMEC 500 µg | Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg | Seq 8: Tiotropium 18 µg, Placebo, UMEC 250 µg, UMEC 500 µg | Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, Placebo | Seq 10: Tiotropium 18 µg, UMEC 250 µg, Placebo, UMEC 500 µg | Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg | Seq 12: UMEC 250 µg, Placebo, UMEC 500 µg, Tiotropium 18 µg
Started | 1 | 4 | 4 | 3 | 3 | 1 | 2 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 4 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Period: Washout Period 1
Arm/Group | Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, Placebo | Seq 2: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg, Placebo | Seq 3: UMEC 250 µg, Placebo, UMEC 500 µg, UMEC 1000 µg | Seq 4: UMEC 250 µg, UMEC 500 µg, Placebo, UMEC 1000 µg | Seq 5: Placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg | Seq 6: UMEC 250 µg, Placebo, Tiotropium 18 µg, UMEC 500 µg | Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg | Seq 8: Tiotropium 18 µg, Placebo, UMEC 250 µg, UMEC 500 µg | Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, Placebo | Seq 10: Tiotropium 18 µg, UMEC 250 µg, Placebo, UMEC 500 µg | Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg | Seq 12: UMEC 250 µg, Placebo, UMEC 500 µg, Tiotropium 18 µg
Started | 1 | 4 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Completed | 1 | 4 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, Placebo | Seq 2: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg, Placebo | Seq 3: UMEC 250 µg, Placebo, UMEC 500 µg, UMEC 1000 µg | Seq 4: UMEC 250 µg, UMEC 500 µg, Placebo, UMEC 1000 µg | Seq 5: Placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg | Seq 6: UMEC 250 µg, Placebo, Tiotropium 18 µg, UMEC 500 µg | Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg | Seq 8: Tiotropium 18 µg, Placebo, UMEC 250 µg, UMEC 500 µg | Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, Placebo | Seq 10: Tiotropium 18 µg, UMEC 250 µg, Placebo, UMEC 500 µg | Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg | Seq 12: UMEC 250 µg, Placebo, UMEC 500 µg, Tiotropium 18 µg
Started | 1 | 4 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Completed | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, Placebo | Seq 2: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg, Placebo | Seq 3: UMEC 250 µg, Placebo, UMEC 500 µg, UMEC 1000 µg | Seq 4: UMEC 250 µg, UMEC 500 µg, Placebo, UMEC 1000 µg | Seq 5: Placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg | Seq 6: UMEC 250 µg, Placebo, Tiotropium 18 µg, UMEC 500 µg | Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg | Seq 8: Tiotropium 18 µg, Placebo, UMEC 250 µg, UMEC 500 µg | Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, Placebo | Seq 10: Tiotropium 18 µg, UMEC 250 µg, Placebo, UMEC 500 µg | Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg | Seq 12: UMEC 250 µg, Placebo, UMEC 500 µg, Tiotropium 18 µg
Started | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Completed | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, Placebo | Seq 2: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg, Placebo | Seq 3: UMEC 250 µg, Placebo, UMEC 500 µg, UMEC 1000 µg | Seq 4: UMEC 250 µg, UMEC 500 µg, Placebo, UMEC 1000 µg | Seq 5: Placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg | Seq 6: UMEC 250 µg, Placebo, Tiotropium 18 µg, UMEC 500 µg | Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg | Seq 8: Tiotropium 18 µg, Placebo, UMEC 250 µg, UMEC 500 µg | Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, Placebo | Seq 10: Tiotropium 18 µg, UMEC 250 µg, Placebo, UMEC 500 µg | Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg | Seq 12: UMEC 250 µg, Placebo, UMEC 500 µg, Tiotropium 18 µg
Started | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Completed | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, Placebo | Seq 2: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg, Placebo | Seq 3: UMEC 250 µg, Placebo, UMEC 500 µg, UMEC 1000 µg | Seq 4: UMEC 250 µg, UMEC 500 µg, Placebo, UMEC 1000 µg | Seq 5: Placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg | Seq 6: UMEC 250 µg, Placebo, Tiotropium 18 µg, UMEC 500 µg | Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg | Seq 8: Tiotropium 18 µg, Placebo, UMEC 250 µg, UMEC 500 µg | Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, Placebo | Seq 10: Tiotropium 18 µg, UMEC 250 µg, Placebo, UMEC 500 µg | Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg | Seq 12: UMEC 250 µg, Placebo, UMEC 500 µg, Tiotropium 18 µg
Started | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Completed | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Seq 1: UMEC 250 µg, UMEC 500 µg, Tiotropium 18 µg, Placebo | Seq 2: UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg, Placebo | Seq 3: UMEC 250 µg, Placebo, UMEC 500 µg, UMEC 1000 µg | Seq 4: UMEC 250 µg, UMEC 500 µg, Placebo, UMEC 1000 µg | Seq 5: Placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg | Seq 6: UMEC 250 µg, Placebo, Tiotropium 18 µg, UMEC 500 µg | Seq 7: Placebo, Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg | Seq 8: Tiotropium 18 µg, Placebo, UMEC 250 µg, UMEC 500 µg | Seq 9: Tiotropium 18 µg, UMEC 250 µg, UMEC 500 µg, Placebo | Seq 10: Tiotropium 18 µg, UMEC 250 µg, Placebo, UMEC 500 µg | Seq 11: Placebo, UMEC 250 µg, Tiotropium 18 µg, UMEC 500 µg | Seq 12: UMEC 250 µg, Placebo, UMEC 500 µg, Tiotropium 18 µg
Started | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Completed | 1 | 3 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Treatments: Participants received a sequence containing 4 of the following 5 possible treatments: placebo, UMEC 250 µg, UMEC 500 µg, UMEC 1000 µg and Tiotropium 18 µg. Participants received each of the treatments in 1 of 4 single dose treatment periods, each of which was followed by a washout period. Treatment periods 1, 2, and 3 were followed by at least a 14-day washout period; Treatment period 4 was followed by a Follow-up visit within 10 days.
Arm/Group | All Study Treatments
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (5.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, or is an event of possible drug-induced liver injury. Refer to the general AE/SAE module for a list of AEs and SAEs.
Time Frame: From Day 1 of Treatment Period 1until Follow-up (up to 10 weeks)
Population: All Subjects Population: all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Groups:
- Placebo: Participants received a single inhaled dose of matching placebo via a dry powder inhaler (DPI) in one of the 4 treatment periods, separated by a washout period of at least 14 days.
- UMEC 250 µg: Participants received a single inhaled dose of a dry powder formulation of UMEC 250 micrograms (µg) via a DPI in one of the 4 treatment periods, separated by a washout period of at least 14 days.
- UMEC 500 µg: Participants received a single inhaled dose of a dry powder formulation of UMEC 500 µg via a DPI in one of the 4 treatment periods, separated by a washout period of at least 14 days.
- UMEC 1000 µg: Participants received a single inhaled dose of a dry powder formulation of UMEC 1000 µg via a DPI in one of the 4 treatment periods, separated by a washout period of at least 14 days.
- Tiotropium 18 µg: Participants received a single inhaled dose of a dry powder formulation of tiotropium 18 µg via a DPI in one of the 4 treatment periods, separated by a washout period of at least 14 days.
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Participants
  Any AE | 6 | 9 | 8 | 4 | 3
  Any SAE | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum (0-4 Hours) Heart Rate on Day 1 of Each Treatment Period
Description: Resting heart rate was measured at pre-dose and 15 minutes (min), 45min, 1.5 hour (h) 4 h, 8 h, and 24 h post-dose of each treatment period and the maximum value for heart rate (0-4hours) was derived at rest. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population. All participants with >=1 post-Baseline assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 1.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute (bpm)
Groups:
- UMEC 250 µg: Participants received a single inhaled dose of a dry powder formulation of UMEC 250 µg via a DPI in one of the 4 treatment periods, separated by a washout period of at least 14 days.
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Beats per minute (bpm) | 69.1 (1.01) | 68.7 (1.14) | 69.5 (1.04) | 71.2 (1.54) | 66.4 (1.69)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-3.0 to 2.2], Standard Error of Mean 1.31
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-2.1 to 2.9], Standard Error of Mean 1.25
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-1.4 to 5.7], Standard Error of Mean 1.77
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-6.2 to 0.9], Standard Error of Mean 1.79
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-1.3 to 5.8], Standard Error of Mean 1.78
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-0.7 to 6.9], Standard Error of Mean 1.89
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-0.1 to 9.7], Standard Error of Mean 2.46

3. Primary Outcome: Weighted Mean (0-4 Hours) Heart Rate at Day 1 of Each Treatment Period
Description: Resting heart rate was measured at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the weighted mean value for heart rate (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Beats per minute (bpm)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Beats per minute (bpm) | 64.66 (0.882) | 63.88 (0.953) | 65.69 (0.894) | 66.61 (1.177) | 62.93 (1.275)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-2.47 to 0.92], Standard Error of Mean 0.844
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.04, 95% CI 2-sided [-0.57 to 2.64], Standard Error of Mean 0.798
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.95, 95% CI 2-sided [-0.35 to 4.26], Standard Error of Mean 1.151
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-4.11 to 0.67], Standard Error of Mean 1.193
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [-1.44 to 3.33], Standard Error of Mean 1.190
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.76, 95% CI 2-sided [0.24 to 5.28], Standard Error of Mean 1.257
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.68, 95% CI 2-sided [0.34 to 7.02], Standard Error of Mean 1.670

4. Primary Outcome: Maximum (0-4 Hours) Systolic Blood Pressure at Day 1 of Each Treatment Period
Description: Resting systolic blood pressure was measured at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the maximum value for systolic blood pressure (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Millimeters of mercury (mmHg) | 129.7 (1.59) | 129.0 (1.84) | 126.2 (1.65) | 133.0 (2.41) | 131.0 (2.78)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-5.0 to 3.4], Standard Error of Mean 2.11
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-7.6 to 0.6], Standard Error of Mean 2.03
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-2.2 to 8.7], Standard Error of Mean 2.74
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-4.7 to 7.2], Standard Error of Mean 2.98
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-7.7 to 3.6], Standard Error of Mean 2.83
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-11.2 to 1.6], Standard Error of Mean 3.20
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-5.9 to 10.0], Standard Error of Mean 4.00

5. Primary Outcome: Weighted Mean (0-4 Hours) Systolic Blood Pressure at Day 1 of Each Treatment Period
Description: Resting systolic blood pressure was measured at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the weighted mean value for systolic blood pressure (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Millimeters of mercury (mmHg) | 124.49 (1.445) | 122.07 (1.670) | 122.61 (1.503) | 125.61 (2.190) | 124.80 (2.517)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.42, 95% CI 2-sided [-6.23 to 1.39], Standard Error of Mean 1.902
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-5.56 to 1.79], Standard Error of Mean 1.834
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-3.82 to 6.07], Standard Error of Mean 2.474
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-5.07 to 5.69], Standard Error of Mean 2.697
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-7.84 to 2.38], Standard Error of Mean 2.562
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.19, 95% CI 2-sided [-7.97 to 3.59], Standard Error of Mean 2.898
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-6.39 to 8.02], Standard Error of Mean 3.618

6. Primary Outcome: Maximum (0-4 Hours) Diastolic Blood Pressure at Day 1 of Each Treatment Period
Description: Resting diastolic blood pressure was measured at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the maximum value for diastolic blood pressure (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Millimeters of mercury (mmHg) | 82.7 (0.96) | 80.2 (1.14) | 80.6 (1.01) | 86.0 (1.46) | 80.3 (1.63)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-5.1 to 0.2], Standard Error of Mean 1.31
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-4.6 to 0.4], Standard Error of Mean 1.25
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-0.0 to 6.6], Standard Error of Mean 1.67
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-5.9 to 1.2], Standard Error of Mean 1.77
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-3.5 to 3.3], Standard Error of Mean 1.71
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-3.5 to 4.1], Standard Error of Mean 1.90
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [1.0 to 10.4], Standard Error of Mean 2.35

7. Primary Outcome: Weighted Mean (0-4 Hours) Diastolic Blood Pressure at Day 1 of Each Treatment Period
Description: Resting diastolic blood pressure was measured at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the weighted mean value for diastolic blood pressure (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Millimeters of mercury (mmHg) | 79.21 (0.759) | 76.23 (0.902) | 77.69 (0.798) | 81.42 (1.156) | 75.89 (1.293)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.97, 95% CI 2-sided [-5.08 to -0.87], Standard Error of Mean 1.051
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-3.53 to 0.50], Standard Error of Mean 1.006
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [-0.46 to 4.88], Standard Error of Mean 1.335
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -3.32, 95% CI 2-sided [-6.13 to -0.50], Standard Error of Mean 1.409
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-2.38 to 3.07], Standard Error of Mean 1.366
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.80, 95% CI 2-sided [-1.22 to 4.82], Standard Error of Mean 1.514
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 5.53, 95% CI 2-sided [1.81 to 9.25], Standard Error of Mean 1.867

8. Primary Outcome: Maximum (0-4 Hours) QTcB at Day 1 of Each Treatment Period
Description: Twelve-lead ECGs (electrocardiograms) were performed to measure QT interval corrected according to Bazzet's formula (QTcB) at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the maximum value for QTcB (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Milliseconds (msec)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Milliseconds (msec) | 402.79 (2.263) | 399.48 (2.621) | 404.48 (2.396) | 401.25 (3.579) | 397.62 (3.867)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -3.31, 95% CI 2-sided [-9.82 to 3.21], Standard Error of Mean 3.256
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.69, 95% CI 2-sided [-4.70 to 8.09], Standard Error of Mean 3.193
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-10.06 to 6.98], Standard Error of Mean 4.268
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -5.17, 95% CI 2-sided [-13.84 to 3.50], Standard Error of Mean 4.347
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.86, 95% CI 2-sided [-6.65 to 10.37], Standard Error of Mean 4.264
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 6.86, 95% CI 2-sided [-2.35 to 16.08], Standard Error of Mean 4.622
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.63, 95% CI 2-sided [-7.59 to 14.85], Standard Error of Mean 5.634

9. Primary Outcome: Weighted Mean (0-4 Hours) QTcB at Day 1 of Each Treatment Period
Description: Twelve-lead ECGs were performed to measure QTcB at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the weighted mean value for QTcB (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Milliseconds (msec)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Milliseconds (msec) | 391.266 (1.7582) | 390.968 (2.0079) | 392.332 (1.8401) | 389.204 (2.7044) | 391.628 (2.9378)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.298, 95% CI 2-sided [-4.961 to 4.365], Standard Error of Mean 2.3297
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.066, 95% CI 2-sided [-3.495 to 5.627], Standard Error of Mean 2.2776
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.062, 95% CI 2-sided [-8.247 to 4.122], Standard Error of Mean 3.0952
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.362, 95% CI 2-sided [-6.003 to 6.726], Standard Error of Mean 3.1891
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.660, 95% CI 2-sided [-6.873 to 5.554], Standard Error of Mean 3.1121
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.704, 95% CI 2-sided [-6.064 to 7.473], Standard Error of Mean 3.3916
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.424, 95% CI 2-sided [-10.84 to 5.993], Standard Error of Mean 4.2233

10. Primary Outcome: Maximum (0-4 Hours) QTcF at Day 1 of Each Treatment Period
Description: Twelve-lead ECGs were performed to measure QT interval corrected according to Fredericia's formula (QTcF) at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the maximum value for QTcF (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Milliseconds (msec)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Milliseconds (msec) | 394.25 (1.699) | 394.34 (1.977) | 395.60 (1.802) | 393.10 (2.604) | 393.93 (2.873)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-4.98 to 5.15], Standard Error of Mean 2.542
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [-3.65 to 6.34], Standard Error of Mean 2.507
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-7.49 to 5.19], Standard Error of Mean 3.182
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-6.89 to 6.24], Standard Error of Mean 3.296
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-6.13 to 6.94], Standard Error of Mean 3.279
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [-5.34 to 8.67], Standard Error of Mean 3.516
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-8.97 to 7.32], Standard Error of Mean 4.087

11. Primary Outcome: Weighted Mean (0-4 Hours) QTcF at Day 1 of Each Treatment Period
Description: Twelve-lead ECGs were performed to measure QTcF at pre-dose and 15 minutes (min), 45 min, 1.5 hours (h), 4 h, 8 h and 24 h post-dose of each treatment period and the weighted mean value for QTcF (0-4 hours) was derived. Baseline is the mean of the 3 pre-dose measurements for each period. Participant level Baseline is the mean of the Baselines for each participant and period level Baseline is the difference between the Baseline and the participant level Baseline in each treatment period for each participant. Analysis was performed using a mixed model with participant level Baseline, period level Baseline, period and treatment group were fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Milliseconds (msec)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Milliseconds (msec) | 386.501 (1.3698) | 387.965 (1.5869) | 386.750 (1.4414) | 383.856 (2.1160) | 389.086 (2.3515)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.464, 95% CI 2-sided [-2.492 to 5.419], Standard Error of Mean 1.9766
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.248, 95% CI 2-sided [-3.647 to 4.144], Standard Error of Mean 1.9457
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.645, 95% CI 2-sided [-7.687 to 2.396], Standard Error of Mean 2.5254
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.585, 95% CI 2-sided [-2.671 to 7.840], Standard Error of Mean 2.6352
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.121, 95% CI 2-sided [-6.308 to 4.067], Standard Error of Mean 2.5993
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.336, 95% CI 2-sided [-7.952 to 3.280], Standard Error of Mean 2.8164
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -5.230, 95% CI 2-sided [-11.96 to 1.504], Standard Error of Mean 3.3802

12. Primary Outcome: Maximum (0-24 Hours) Heart Rate as Measured From Holter Monitoring at Day 1 of Each Treatment Period
Description: Twenty-four hour Holter monitoring was conducted to measure heart rate for the 24-hour period following dosing at each treatment period and the maximum value for heart rate (0-24 hours) was derived. Analysis was performed using a mixed model of period and treatment group fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Beats per minute (bpm)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Beats per minute (bpm) | 116.7 (2.92) | 111.5 (3.06) | 112.1 (2.96) | 109.0 (3.53) | 111.4 (3.79)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-9.7 to -0.7], Standard Error of Mean 2.24
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-8.9 to -0.3], Standard Error of Mean 2.15
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-13.5 to -1.8], Standard Error of Mean 2.91
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-11.8 to 1.1], Standard Error of Mean 3.21
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-6.1 to 6.4], Standard Error of Mean 3.12
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-6.1 to 7.5], Standard Error of Mean 3.38
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-10.9 to 6.2], Standard Error of Mean 4.29

13. Primary Outcome: Mean (0-24 Hours) Heart Rate as Measured From Holter Monitoring at Day 1 of Each Treatment Period
Description: Twenty-four-hour Holter monitoring was conducted to measure heart rate for the 24-h period following dosing of each treatment period and the mean value for heart rate (0-24 hours) was derived. Analysis was performed using a mixed model of period and treatment group fitted as fixed effects and participant as a random effect.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Beats per minute (bpm)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Beats per minute (bpm) | 77.1 (1.61) | 75.3 (1.66) | 76.8 (1.62) | 75.5 (1.80) | 76.1 (1.89)
Statistical Analysis 1: Comparison: Placebo vs UMEC 250 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.6 to 0.0], Standard Error of Mean 0.90
Statistical Analysis 2: Comparison: Placebo vs UMEC 500 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.0 to 1.4], Standard Error of Mean 0.86
Statistical Analysis 3: Comparison: Placebo vs UMEC 1000 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.9 to 0.8], Standard Error of Mean 1.17
Statistical Analysis 4: Comparison: Placebo vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-3.6 to 1.6], Standard Error of Mean 1.30
Statistical Analysis 5: Comparison: UMEC 250 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-3.3 to 1.7], Standard Error of Mean 1.26
Statistical Analysis 6: Comparison: UMEC 500 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-2.0 to 3.4], Standard Error of Mean 1.37
Statistical Analysis 7: Comparison: UMEC 1000 µg vs Tiotropium 18 µg; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-4.1 to 2.9], Standard Error of Mean 1.74

14. Primary Outcome: Basophils, Eosinophils, Lymphocytes, Monocytes, and Total Neutrophils Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, and total neutrophils at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Percentage
  Basophils, Pre-dose | 0.65 (0.284) | 0.73 (0.366) | 0.74 (0.396) | 0.87 (0.275) | 0.71 (0.314)
  Basophils, 24 h Post-dose | 0.70 (0.434) | 0.65 (0.313) | 0.56 (0.292) | 0.58 (0.344) | 0.76 (0.558)
  Eosinophils, Pre-dose | 3.30 (2.336) | 3.46 (2.249) | 3.67 (2.813) | 4.03 (2.679) | 3.05 (1.562)
  Eosinophils, 24 h Post-dose | 3.34 (1.914) | 3.25 (1.839) | 3.30 (2.164) | 3.49 (2.437) | 3.38 (1.552)
  Lymphocytes, Pre-dose | 29.23 (6.820) | 30.66 (7.355) | 28.91 (9.279) | 33.70 (7.161) | 27.99 (7.637)
  Lymphocytes, 24 h Post-dose | 31.60 (6.387) | 30.86 (6.749) | 30.99 (6.558) | 31.72 (4.920) | 30.86 (6.298)
  Monocytes, Pre-dose | 8.53 (1.842) | 8.50 (2.467) | 8.60 (2.179) | 8.10 (1.626) | 9.33 (2.582)
  Monocytes, 24 h Post-dose | 8.10 (1.975) | 7.62 (1.934) | 8.23 (1.985) | 7.45 (1.406) | 9.40 (2.084)
  Total neutrophils, Pre-dose | 58.30 (8.159) | 56.64 (9.081) | 58.10 (10.941) | 53.32 (7.825) | 58.88 (9.403)
  Total neutrophils, 24 h Post-dose | 56.26 (7.166) | 57.62 (7.740) | 56.94 (7.164) | 56.78 (6.204) | 55.63 (7.699)

15. Primary Outcome: Hemoglobin, Mean Corpuscle Hemoglobin Concentration (MCHC), Albumin and Total Protein Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of hemoglobin, MCHC, albumin and total protein at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Grams per liter (G/L)
  Hemoglobin, Pre-dose | 146.1 (11.80) | 146.6 (10.31) | 145.4 (11.27) | 143.8 (12.34) | 152.0 (7.23)
  Hemoglobin, 24 h Post-dose | 147.0 (12.53) | 145.5 (11.01) | 144.1 (10.97) | 143.5 (14.77) | 148.9 (5.59)
  MCHC, Pre-dose | 347.2 (7.03) | 343.3 (5.78) | 344.1 (7.87) | 346.8 (4.62) | 343.0 (5.04)
  MCHC, 24 h Post-dose | 344.9 (6.35) | 344.0 (7.02) | 344.9 (8.50) | 345.2 (6.57) | 342.9 (3.91)
  Albumin, Pre-dose | 39.16 (2.020) | 39.24 (2.109) | 39.33 (1.955) | 39.10 (1.545) | 39.49 (2.775)
  Albumin, 24 h Post-dose | 39.36 (1.682) | 38.75 (1.742) | 38.76 (1.744) | 39.30 (1.750) | 38.38 (2.930)
  Total protein, Pre-dose | 66.05 (4.120) | 66.04 (4.245) | 66.19 (3.987) | 66.15 (3.576) | 65.35 (2.931)
  Total protein, 24 h Post-dose | 66.37 (3.584) | 65.40 (3.933) | 65.62 (2.945) | 66.44 (3.448) | 64.14 (3.349)

16. Primary Outcome: Hematocrit Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of hematocrit at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Proportion of red blood cells in blood
  Pre-dose | 0.421 (0.0335) | 0.428 (0.0321) | 0.423 (0.0326) | 0.416 (0.0345) | 0.445 (0.0193)
  24 h Post-dose | 0.427 (0.0352) | 0.424 (0.0361) | 0.418 (0.0322) | 0.417 (0.0419) | 0.434 (0.0192)

17. Primary Outcome: Mean Corpuscle Hemoglobin Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of the mean corpuscle hemoglobin at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: picograms/cell (pg)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
picograms/cell (pg)
  Pre-dose | 32.56 (1.402) | 32.36 (1.365) | 32.36 (1.513) | 32.29 (1.393) | 32.86 (0.971)
  24 Hour Post-dose | 32.41 (1.354) | 32.36 (1.208) | 32.36 (1.359) | 32.15 (1.309) | 32.79 (1.018)

18. Primary Outcome: Mean Corpuscle Volume Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of the mean corpuscle volume at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Femtoliters (FL)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Femtoliters (FL)
  Pre-dose | 93.78 (3.701) | 94.23 (3.547) | 94.04 (3.734) | 93.11 (3.840) | 95.83 (3.310)
  24 h Post-dose | 93.99 (3.597) | 94.09 (3.763) | 93.85 (3.955) | 93.15 (3.652) | 95.65 (2.946)

19. Primary Outcome: Red Blood Cells Count Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of the red blood cells count at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
10^12 cells per liter (TI/L)
  Pre-dose | 4.493 (0.3992) | 4.537 (0.3487) | 4.498 (0.3758) | 4.456 (0.3987) | 4.625 (0.2469)
  24 h Post-dose | 4.539 (0.3960) | 4.498 (0.3760) | 4.457 (0.3614) | 4.464 (0.4511) | 4.543 (0.2232)

20. Primary Outcome: Platelets Count and White Blood Cells (WBC) Count Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of platelets count and WBC count at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
10^9 cells per liter (GI/L)
  Platelets count, Pre-dose | 247.2 (70.84) | 245.0 (71.33) | 250.7 (69.06) | 235.9 (47.15) | 243.4 (104.43)
  Platelets count, 24 h Post-dose | 248.8 (69.53) | 245.4 (76.18) | 250.3 (63.51) | 237.9 (46.30) | 237.6 (101.59)
  WBC count, Pre-dose | 7.623 (1.7271) | 7.130 (1.6116) | 7.560 (1.6860) | 7.121 (1.2807) | 6.763 (1.0249)
  WBC count, 24 h Post-dose | 7.520 (1.3103) | 7.385 (1.7548) | 7.218 (1.4426) | 7.999 (1.6531) | 6.623 (1.2366)

21. Primary Outcome: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Phosphokinase (CPK), and Gamma Glutamyl Transferase (GGT) Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of ALP, ALT, AST, CPK, and GGT at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles). Different participants may have been summarized for different parameters/at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
International units per liter (IU/L)
  ALP, Pre-dose, n=21, 22, 21, 13, 8 | 67.04 (17.260) | 65.32 (12.687) | 66.60 (13.127) | 63.37 (13.469) | 71.06 (19.304)
  ALP, 24 h Post-dose, n=21, 22, 21, 13, 8 | 67.20 (18.388) | 65.04 (15.289) | 64.96 (14.933) | 61.76 (12.253) | 71.84 (21.099)
  ALT, Pre-dose,n=21, 22, 21, 13, 8 | 23.6 (11.67) | 24.1 (9.80) | 21.3 (8.37) | 26.2 (10.53) | 19.1 (5.36)
  ALT, 24 h Post-dose,n=21, 22, 21, 13, 8 | 23.3 (12.29) | 23.0 (9.36) | 20.5 (7.56) | 25.6 (9.69) | 17.8 (5.39)
  AST, Pre-dose, n=21, 22, 20, 13, 8 | 21.98 (7.525) | 24.55 (6.689) | 22.13 (5.358) | 23.03 (6.923) | 22.09 (4.995)
  AST, 24 h Post-dose, n=21, 22, 21, 13, 8 | 21.68 (8.625) | 22.01 (7.048) | 20.58 (5.761) | 20.75 (6.947) | 19.23 (5.473)
  CPK, Pre-dose, n=21, 22, 21, 13, 8 | 124.33 (89.568) | 101.88 (49.410) | 104.39 (42.381) | 100.16 (44.497) | 117.08 (61.189)
  CPK, 24 h Post-dose, n=21, 22, 21, 13, 8 | 99.97 (61.307) | 82.81 (30.913) | 83.77 (29.233) | 87.78 (37.566) | 109.36 (90.411)
  GGT, Pre-dose, n=21, 22, 21, 13, 8 | 27.81 (18.287) | 26.41 (14.704) | 26.41 (17.573) | 29.86 (21.391) | 19.94 (6.369)
  GGT, 24 h Post-dose, n=21, 22, 21, 13, 8 | 27.14 (16.806) | 25.33 (13.962) | 25.89 (18.218) | 29.38 (19.277) | 19.59 (6.431)

22. Primary Outcome: Total Bilirubin, Creatinine and Uric Acid Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of total bilirubin, creatinine, and uric acid at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Micromoles per liter (µmol/L)
  Total bilirubin, Pre-dose | 7.92 (2.457) | 8.33 (2.234) | 8.66 (3.387) | 8.68 (2.238) | 7.69 (1.549)
  Total bilirubin, 24 h Post-dose | 8.70 (2.602) | 8.26 (2.955) | 9.48 (3.523) | 10.27 (3.086) | 6.83 (2.036)
  Creatinine, Pre-dose | 78.55 (7.589) | 80.50 (8.012) | 80.24 (10.079) | 78.64 (8.296) | 79.79 (8.333)
  Creatinine, 24 h Post-dose | 78.02 (6.451) | 79.08 (8.324) | 78.14 (9.684) | 76.44 (7.241) | 76.29 (8.999)
  Uric acid, Pre-dose | 295.86 (64.155) | 301.24 (77.192) | 303.18 (77.389) | 317.09 (76.125) | 281.19 (67.657)
  Uric acid, 24 h Post-dose | 285.55 (63.350) | 293.21 (65.637) | 296.28 (70.307) | 306.26 (72.701) | 268.64 (61.525)

23. Primary Outcome: Calcium, Bicarbonate, Chloride, Glucose, Inorganic Phosphorus (IP), Potassium, Sodium, and Urea Values at the Indicated Time Points on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of the calcium, bicarbonate, chloride, glucose, IP, potassium, sodium, and urea at pre-dose and 24 hour (h) post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles). Different participants may have been analyzed for different parameters/at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Millimoles per liter (mmol/L)
  Calcium, Pre-dose, n=21, 22, 21, 13, 8 | 2.283 (0.0729) | 2.277 (0.0861) | 2.267 (0.0809) | 2.242 (0.0625) | 2.278 (0.0547)
  Calcium, 24 h Post-dose, n=21, 22, 21, 13, 8 | 2.270 (0.0891) | 2.290 (0.0713) | 2.265 (0.0704) | 2.244 (0.0864) | 2.280 (0.0428)
  Chloride, Pre-dose, n=21, 22, 21, 13, 8 | 106.88 (2.727) | 107.11 (1.972) | 106.42 (1.857) | 107.26 (2.738) | 106.49 (2.255)
  Chloride, 24 h Post-dose, n=21, 22, 21, 13, 8 | 107.18 (1.875) | 107.10 (2.457) | 106.94 (2.002) | 107.17 (2.830) | 106.59 (1.460)
  Glucose, Pre-dose, n=21, 22, 21, 13, 8 | 5.225 (0.5294) | 5.046 (0.5583) | 5.082 (0.5882) | 5.098 (0.4362) | 5.326 (0.6739)
  Glucose, 24 h Post-dose, n=21, 22, 21, 13, 8 | 5.278 (0.5800) | 5.203 (0.6391) | 5.224 (0.5500) | 5.031 (0.3691) | 5.291 (0.5350)
  Bicarbonate, Pre-dose, n=21, 22, 21, 13, 8 | 22.41 (2.609) | 22.95 (2.295) | 23.28 (2.698) | 23.08 (2.401) | 22.98 (4.179)
  Bicarbonate, 24 h Post-dose, n=21, 22, 21, 13, 7 | 22.98 (2.414) | 22.62 (2.995) | 23.30 (2.600) | 23.80 (2.822) | 25.14 (2.738)
  Potassium, Pre-dose, n=21, 22, 21, 13, 8 | 4.283 (0.3178) | 4.177 (0.2537) | 4.209 (0.2255) | 4.248 (0.2717) | 4.193 (0.1896)
  Potassium, 24 h Post-dose, n=21, 22, 21, 13, 8 | 4.270 (0.2340) | 4.274 (0.3311) | 4.266 (0.3065) | 4.279 (0.3587) | 4.359 (0.3642)
  Sodium, Pre-dose,n=21, 22, 21, 13, 8 | 140.45 (2.253) | 140.95 (1.932) | 140.84 (1.551) | 141.07 (0.825) | 140.86 (2.458)
  Sodium, 24 h Post-dose, n=21, 22, 21, 13, 8 | 140.90 (1.674) | 140.68 (1.864) | 140.93 (1.610) | 141.13 (1.165) | 140.56 (1.749)
  IP, Pre-dose, n=21, 22, 21, 13, 8 | 1.153 (0.1271) | 1.095 (0.1026) | 1.135 (0.1406) | 1.105 (0.1490) | 1.161 (0.1763)
  IP, 24 h Post-dose, n=21, 22, 21, 13, 8 | 1.131 (0.1455) | 1.118 (0.1391) | 1.143 (0.1486) | 1.121 (0.1735) | 1.158 (0.1179)
  Urea, Pre-dose, n=21, 22, 21, 13, 8 | 4.905 (1.2041) | 4.629 (0.9289) | 5.002 (1.1933) | 4.904 (0.9358) | 4.820 (1.2474)
  Urea, 24 h Post-dose, n=21, 22, 21, 13, 8 | 4.700 (0.8093) | 4.721 (0.9688) | 4.710 (0.9958) | 4.579 (0.8701) | 4.764 (1.6021)

24. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) at the Indicated Time Points on Day 1 of Each Treatment Period
Description: FEV1 and FVC are measures of lung function. FEV1 is defined as the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. FEV1 and FVC measurements were taken at pre-dose and 1 hour (h), 2 h, 6 h, 9 h, 12 h and 24 h post-dose of each treatment period.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Liters
  FEV1, Pre-dose, n= 21, 22, 21, 13, 8 | 1.637 (0.3991) | 1.559 (0.2867) | 1.589 (0.2871) | 1.732 (0.2080) | 1.400 (0.2545)
  FEV1, 1h, n=21, 20, 21, 13, 8 | 1.670 (0.4130) | 1.874 (0.3414) | 1.905 (0.3574) | 1.966 (0.3781) | 1.663 (0.3250)
  FEV1, 2h, n= 21, 20, 21, 13, 8 | 1.689 (0.4172) | 1.969 (0.3760) | 2.015 (0.3512) | 2.123 (0.3757) | 1.696 (0.3311)
  FEV1, 6h, n=21, 22, 21, 13, 8 | 1.700 (0.4055) | 2.000 (0.4251) | 2.073 (0.3343) | 2.198 (0.3329) | 1.841 (0.4372)
  FEV1, 9h, n=21, 19, 21, 13, 7 | 1.754 (0.3664) | 1.984 (0.3554) | 2.010 (0.3113) | 2.135 (0.2850) | 1.767 (0.4555)
  FEV1, 12h, n=21, 22, 21, 13,8 | 1.688 (0.3797) | 1.933 (0.3756) | 1.988 (0.3463) | 2.103 (0.3633) | 1.619 (0.4182)
  FEV1, 24h, =21, 22, 21, 13, 8 | 1.612 (0.3189) | 1.830 (0.4033) | 1.817 (0.3569) | 1.978 (0.3416) | 1.454 (0.3135)
  FVC, Pre-dose, n=21, 22, 21, 13, 8 | 3.438 (0.8138) | 3.247 (0.7574) | 3.337 (0.7139) | 3.640 (0.7869) | 3.080 (0.6682)
  FVC, 1h, n=21, 20, 21, 13, 8 | 3.490 (0.8721) | 3.751 (0.8688) | 3.845 (0.7974) | 4.006 (0.9430) | 3.631 (0.7223)
  FVC, 2h, n=21, 20, 21, 13, 8 | 3.545 (0.8796) | 3.877 (0.9571) | 3.976 (0.8479) | 4.205 (0.9935) | 3.674 (0.7766)
  FVC, 6h, n=21, 22, 21, 13, 8 | 3.572 (0.8555) | 3.940 (0.9583) | 4.064 (0.8822) | 4.257 (1.0390) | 3.780 (0.8023)
  FVC, 9h, n=21, 19, 21, 13, 7 | 3.662 (0.8436) | 4.015 (0.8461) | 3.969 (0.8783) | 4.184 (0.9694) | 3.544 (0.7176)
  FVC, 12h, n=21, 22, 21, 13, 8 | 3.595 (0.8178) | 3.841 (0.9190) | 3.923 (0.8966) | 4.130 (1.0544) | 3.563 (0.7816)
  FVC, 24h, n=21, 22, 21, 13, 8 | 3.389 (0.7272) | 3.712 (0.9878) | 3.705 (0.8597) | 3.993 (0.9759) | 3.280 (0.6741)

25. Secondary Outcome: Area Under Concentration-time Curve From Time 0 to 2 Hours [AUC(0-2)] and Area Under Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration [AUC(0-t)] of UMEC
Description: Blood samples were collected to determine the plasma concentrations of UMEC from pre-dose up to 24 hour post-dose of each treatment period to derive the AUC(0-2) and AUC(0-t). Blood samples for PK analysis of UMEC were obtained on Day 1at pre-dose and 5 minutes (min), 15 min, 30 min, 1 hour (h), 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, and 24 h post UMEC dose administration.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: Pharmacokinetic (PK) Population:all participants in the All Subjects Population for whom a PK sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr * nanograms per milliliter (ng/mL)
Arm/Group | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg
Number analyzed (Participants) | 22 | 21 | 13
hr * nanograms per milliliter (ng/mL)
  AUC(0-2) | 0.10264 (58.9) | 0.27099 (58.5) | 0.71522 (21.8)
  AUC(0-t) | 0.10271 (70.0) | 0.35491 (65.2) | 0.96100 (27.7)

26. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of UMEC
Description: Blood samples were collected to determine the plasma concentrations of UMEC from pre-dose up to 24 hour post-dose of each treatment period to derive the Cmax. Blood samples for PK analysis of UMEC were obtained on Day 1at pre-dose and 5 minutes (min), 15 min, 30 min, 1 hour (h), 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, and 24 h post UMEC dose administration.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg
Number analyzed (Participants) | 22 | 21 | 13
ng/mL | 0.12615 (43.4) | 0.30389 (40.7) | 0.83228 (22.9)

27. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax), Last Time Point Where the Concentration is Above the Limit of Quantification (Tlast), and Plasma Half-life (t1/2) of UMEC
Description: Blood samples were collected to determine the plasma concentrations of UMEC from pre-dose up to 24 hour post-dose of each treatment period to derive tmax, tlast and t1/2. Blood samples for PK analysis of UMEC were obtained on Day 1at pre-dose and 5 minutes (min), 15 min, 30 min, 1 hour (h), 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, and 24 h post UMEC dose administration.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: PK Population. Only those participants with non-missing observations (including non-calculable values) were analyzed (represented by n=X, X, X in the category titles). Different participants may have been analyzed for different parameters/at different time points, so the overall number of participants analyzed reflects everyone in the PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg
Number analyzed (Participants) | 22 | 21 | 13
Hours
  tmax, n=22, 21, 13 | 0.090 [0.08 to 0.50] | 0.100 [0.07 to 0.27] | 0.250 [0.08 to 0.28]
  tlast, n=22, 21, 13 | 1.975 [0.47 to 4.07] | 4.030 [1.00 to 24.00] | 6.000 [4.00 to 15.95]
  t1/2, n=22, 21, 13 | NA [NA to NA] — Due to the large amount of non-quantifiable (NQ) data in the distribution and elimination phase at 250mcg dose level, all t½ values could not be calculated and median and the confidence interval (CI) could not be estimated. | 1.24490 [0.7079 to 3.6743] | 1.19780 [0.7889 to 20.2309]

28. Secondary Outcome: Amount of Drug Excreted Unchanged in Urine From Time Zero to: 2h [Ae(0-2)] , 8h [Ae(0-8)], 12h [Ae(0-12)], 24h [Ae(0-24)], and 48h [Ae(0-48)]; and Area Under the Excretion Rate Curve From Time Zero to: 18h [AUER(0-18)] and 36h [AUER(0-36)] for UMEC
Description: Urine samples were collected to determine the urine concentrations of UMEC from 0 min up to 48 hours post-dose of each treatment period to derive Ae(0-2), Ae(0-8), Ae(0-12), Ae(0-24), Ae(0-48), AUER(0-18) and AUER(0-36). Urine samples for PK analysis of UMEC were obtained on Day 1; a single sample was collected at each of the following timepoints: 0-2 h, 2-8 h, 8-12 h, 12-24 h and 24-48 h post UMEC dose administration.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg
Number analyzed (Participants) | 22 | 21 | 13
ng
  Ae(0-2) | 734.525 (56.0) | 1793.951 (40.5) | 4456.582 (43.5)
  Ae(0-8) | 1676.101 (54.7) | 4146.206 (50.6) | 9935.792 (33.4)
  Ae(0-12) | 1987.910 (50.0) | 4712.376 (50.1) | 10983.771 (34.5)
  Ae(0-24) | 2352.662 (47.5) | 5486.724 (48.3) | 12401.722 (33.7)
  Ae(0-48) | 2729.434 (45.0) | 6361.233 (47.0) | 13671.981 (34.7)
  AUER(0-18) | 2119.916 (48.4) | 4830.401 (47.9) | 10919.838 (34.6)
  AUER(0-36) | 2487.288 (48.8) | 5752.880 (49.3) | 12363.246 (35.0)

29. Secondary Outcome: Renal Clearance (CLr) of UMEC Following Dose Administration on Day 1
Description: The CLr is defined as the apparent total clearance of the drug from plasma after oral administration. Blood samples for PK analysis of UMEC were obtained on Day 1at pre-dose and 5 minutes (min), 15 min, 30 min, 1 hour (h), 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, and 24 h post UMEC dose administration.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/hr)
Arm/Group | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg
Number analyzed (Participants) | 22 | 21 | 13
Liters per hour (L/hr) | 5.317 (56.2) | 6.395 (36.9) | 6.831 (56.8)

30. Secondary Outcome: Half-life for Renal Excretion of UMEC on Day 1
Description: The terminal half-life (t1/2) of UMEC is defined as the time required for the urine concentration of UMEC to reach half of its original concentration. Urine samples for PK analysis of UMEC were obtained on Day 1; a single sample was collected at each of the following timepoints: 0-2 h, 2-8 h, 8-12 h, 12-24 h and 24-48 h post UMEC dose administration.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg
Number analyzed (Participants) | 22 | 21 | 13
Hours | 10.679 (37.2) | 12.023 (44.9) | 10.821 (32.8)

31. Secondary Outcome: Fraction of Dose Excreted Unchanged in Urine From Time Zero to: 24 Hours [Fe(0-24)] and 48 Hours [Fe(0-48)] for UMEC
Description: Urine samples were collected to determine the urine concentrations of UMEC from 0 min up to 48 hours post-dose of each treatment period to derive Fe(0-24) and Fe(0-48). Urine samples for PK analysis of UMEC were obtained on Day 1; a single sample was collected at each of the following timepoints: 0-2 h, 2-8 h, 8-12 h, 12-24 h and 24-48 h post UMEC dose administration.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: PK Population
Measure: Median (Full Range); unit: Percentage of total dose administered
Arm/Group | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg
Number analyzed (Participants) | 22 | 21 | 13
Percentage of total dose administered
  Fe(0-24) | 0.993 [0.32 to 2.56] | 1.253 [0.46 to 2.73] | 1.360 [0.68 to 1.94]
  Fe(0-48) | 1.142 [0.42 to 2.88] | 1.413 [0.48 to 2.95] | 1.512 [0.77 to 2.10]

32. Secondary Outcome: Mean Serial FEV1over 24 Hours After Dosing on Day 1 of Each Treatment Period
Description: Serial spirometry assessments were conducted on Day 1 of each treatment period over the course of 24 hours and were taken at 1 hour (h), 2 h, 6 h, 9 h, 12 h and 24 h post-dose. The maximum of the 3 FEV1 measurements for each participant, treatment period and timepoint were used in the calculation of the mean for each treatment group at each timepoint.
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
Liters
  FEV1, 1 h, n= 21, 20, 21, 13, 8 | 1.638 (0.0410) | 1.861 (0.0437) | 1.915 (0.0408) | 1.834 (0.0542) | 1.880 (0.0644)
  FEV1, 2h, n= 21, 20, 21, 13, 8 | 1.654 (0.0433) | 1.951 (0.0456) | 2.027 (0.0431) | 1.992 (0.0570) | 1.910 (0.0684)
  FEV1, 6h, n=21, 22, 21, 13, 8 | 1.669 (0.0497) | 1.991 (0.0510) | 2.083 (0.0492) | 2.070 (0.0648) | 2.050 (0.0793)
  FEV1, 9h, n=21, 19, 21, 13, 7 | 1.721 (0.0418) | 1.938 (0.0446) | 2.021 (0.0416) | 2.024 (0.0553) | 1.927 (0.0673)
  FEV1, 12h, n=21, 22, 21, 13, 7 | 1.662 (0.0501) | 1.917 (0.0514) | 1.996 (0.0497) | 1.988 (0.0654) | 1.812 (0.0801)
  FEV1, 24h, n=21, 22, 21, 13, 8 | 1.583 (0.0411) | 1.818 (0.0431) | 1.827 (0.0410) | 1.856 (0.0544) | 1.655 (0.0646)

33. Secondary Outcome: Mean Serial Specific Airway Resistance (sGaw) Over 24 Hours After Dosing on Day 1 of Each Treatment Period
Description: sGaw is the specific airways resistance (mid) which was assessed by whole body plethysmography. Values used were the mean of the 3 readings recorded at each timepoint. sGaw measurements were taken at 2 hour (h), 6 h, 12 h and 24 h post-dose of each treatment period. 1/kPa.s=1(the inverses)/kPa (kilopascal).s (second)
Time Frame: Day 1 of each treatment period (up to Study Day 46)
Population: as for outcome 21
Measure: Geometric Mean (Standard Error); unit: 1/kPa*s
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Number analyzed (Participants) | 21 | 22 | 21 | 13 | 8
1/kPa*s
  sGaw, 2h, n= 21, 20, 21, 13, 8 | 0.400 (0.0598) | 0.652 (0.0631) | 0.699 (0.0602) | 0.714 (0.0753) | 0.648 (0.0893)
  sGaw, 6h, n=21, 21, 21, 13, 8 | 0.426 (0.0574) | 0.734 (0.0603) | 0.806 (0.0578) | 0.778 (0.0720) | 0.711 (0.0848)
  sGaw, 12h, n=21, 21, 21, 13, 8 | 0.403 (0.0661) | 0.637 (0.0692) | 0.735 (0.0665) | 0.730 (0.0836) | 0.550 (0.1008)
  sGaw, 24h, n=21, 21, 21, 13, 8 | 0.379 (0.0627) | 0.514 (0.0662) | 0.501 (0.0630) | 0.514 (0.0790) | 0.440 (0.0945)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from Day 1 of Treatment Period 1 until Follow-up visit (up to 10 weeks)
Description: AEs and SAEs were collected in the members of All Subjects Population comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | UMEC 250 µg | UMEC 500 µg | UMEC 1000 µg | Tiotropium 18 µg
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/21 | 0/13 | 0/8
Other Adverse Events (participants affected / at risk) | 6/21 | 9/22 | 8/21 | 4/13 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | UMEC 250 µg (N=22) | UMEC 500 µg (N=21) | UMEC 1000 µg (N=13) | Tiotropium 18 µg (N=8)
Headache (Nervous system disorders) | 4 | 4 | 4 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Infected insect bite (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.